CLINICAL TRIAL: NCT06266299
Title: A Phase 1, Multicenter, Open-label, Dose-escalation Study Evaluating the Safety and Tolerability of Intravenous KK2269 Monotherapy and Combination Therapy With Docetaxel in Adult Participants With Solid Tumors
Brief Title: A Study of KK2269 in Adult Participants With Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2269-001
Record Dates: First submitted 2024-02-05; First posted 2024-02-20 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma; Non Small Cell Lung Cancer
MeSH Terms: conditions — Neoplasm Metastasis; Adenocarcinoma Of Esophagus; Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1 (Experimental): KK2269 will be administered at each dose level, intravenous infusion.
  Interventions: Drug: KK2269
- Part 2 (Experimental): KK2269 will be administered at each dose level intravenously in combination with docetaxel.
  Docetaxel will be administered intravenously (Q3W).
  Interventions: Drug: KK2269; Drug: Docetaxel

INTERVENTIONS:
Drug: KK2269 — KK2269 administered intravenously
Drug: Docetaxel — antineoplastic drug administered intravenously
  Other Names: Docetaxel Hydrate
  Arms: Part 2

SUMMARY:
This is a first-in-human study of KK2269. Part 1 and Part 2 will be conducted as a multicenter, open-label, non-randomized, dose-escalation study. Participants with advanced or metastatic solid tumors for which no standard therapy is available will be enrolled in Part 1. In Part 1, the primary objective is to assess the safety and tolerability of KK2269.

In Part 2, only participants with gastric adenocarcinoma, GEJ adenocarcinoma, esophageal adenocarcinoma, or NSCLC who have experienced at least one systemic therapy will be enrolled. In Part 2, the primary objective is to assess the safety and tolerability of KK2269 in combination with docetaxel and to determine the recommended dose(s) and dose interval(s) of KK2269 in combination with docetaxel for subsequent studies.

In both Part 1 and Part 2, participants who refuse to undergo standard therapy are also eligible.

ELIGIBILITY:
* Key Common Inclusion Criteria for Parts 1 and 2:

  * Patients who are ≥ 18 years old at the time of informed consent
  * Patients who have disease measurable by RECIST v1.1
  * Patients with an ECOG PS of 0 or 1
  * Patients with a life expectancy of at least 3 months in the judgement of the investigator or subinvestigator
  * The specified periods have passed respectively after the completion of previous cancer treatments as of the date of enrollment at the time of the first dose of KK2269
  * Patients who agree to use a medically effective method of contraception
* Key Additional Inclusion Criterion for Part 1:

  •Patients with histological or cytological evidence of at least one locally advanced or metastatic non-CNS solid tumor
* Key Additional Inclusion Criteria for Part 2:

  •Patients with histological or cytological evidence of any of the following disease: Gastric adenocarcinoma, GEJ adenocarcinoma, or esophageal adenocarcinoma, NSCLC (Only patients with NSCLC will be enrolled in the expansion part)

  •Patients who are suitable for docetaxel treatment
* Key Common Exclusion Criteria for Parts 1 and 2:

  * Patients with an uncontrolled or serious intercurrent illness
  * Patients with known active central nervous system metastasis
  * Patients with a history of ≥ Grade 3 allergic reaction to any antibody drug
  * Patients with a history of autoimmune disease
  * Patients with a history of HIV, HBV, or HCV at screening
  * Patients who have a history of primary immunodeficiency
* Key Additional Exclusion Criterion For Part 2:

  * Patients with a history of treatment with docetaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects Experiencing Dose-limiting Toxicity | 21 days after first dose
Number of Adverse Events | From signing of ICF through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - City Of Hope National Medical Center, Duarte, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Washington University, St Louis, Missouri
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Washington, Seattle, Washington
- Japan (4):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Cancer Institute Hospital of JFCR, Koto-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated and/or analyzed during the study sponsored by Kyowa Kirin will be available in the Vivli repository, https://vivli.org/ourmember/kyowa-kirin/ as long as conditions of data disclosure specified in the policy section of the Vivli website are satisfied.
URL: https://vivli.org/ourmember/kyowa-kirin/